CLINICAL TRIAL: NCT04062760
Title: Safety and Efficacy of Early, seQUential Oral dIuretic Nephron blockAde In Acute Heart Failure (SEEQUOIA-AHF)
Brief Title: Safety and Efficacy of Early, seQUential Oral dIuretic Nephron blockAde In Acute Heart Failure
Acronym: SEEQUOIA-AHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other); Azienda USL di Parma (Unknown); Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, Enrico Fiaccadori, Associate Professor of Nephrology, University of Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEEQUOIA-AHF
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Acute Heart Failure
Keywords: Acute Heart Failure; Diuretics; Sequential nephron blockade; Fluid balance; Worsening kidney failure

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, open-label, parallel-arm trial. Eligible patients will be randomized in a 1:1 proportion to treatment with either high-dose oral furosemide or sequential nephron blockade with different classes of diuretics at low doses.
  The primary endpoint will be the bivariate change in body weight and serum creatinine value at 96 hours since patient randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard diuretic therapy (SDT) (Active Comparator): Furosemide +/- spironolactone or potassium canrenoate
  Interventions: Drug: Standard diuretic therapy
- Early sequential nephron blockade (ESNB) (Experimental): Furosemide + metolazone + acetazolamide +/- spironolactone or potassium canrenoate
  Interventions: Drug: Early sequential nephron blockade

INTERVENTIONS:
Drug: Standard diuretic therapy — The patients in this arm will be randomized to receiving oral furosemide in 2 daily divided doses at twice the intravenous dose administered during the past 24 hours. Unless serum potassium value is higher than 5 mmol/L, oral spironolactone or potassium canrenoate will be added; dose will be established based on serum creatinine value.
  Arms: Standard diuretic therapy (SDT)
Drug: Early sequential nephron blockade — After 24-72 hours of an algorithm-based treatment with high-dose intravenous furosemide started at the time of hospital admission, the patients in this arm will be randomized to receiving:
  1. oral furosemide in 2 daily divided doses at a dose equivalent to that administered intravenously during the past 24 hours
  2. metolazone at a dose based on serum creatinine value
  3. acetazolamide at a dose based on serum creatinine value
  4. spironolactone or potassium canrenoate (unless serum potassium value is higher than 5 mmol/L); dose will be established based on serum creatinine value
  Arms: Early sequential nephron blockade (ESNB)

SUMMARY:
The SEEQUOIA-AHF (Safety and Efficacy of Early, seQUential oral dIuretic nephron blockAde in Acute Heart Failure) trial is a multicenter, randomized, open-label, parallel-arm trial assessing the impact of early sequential nephron blockade (i.e. a regimen based on the combination of four oral diuretics with different sites of action along the nephron at low doses) compared to a conventional approach with a high-dose loop diuretic in the treatment of congestion in patients hospitalized with acute heart failure (AHF).

In this study, after 24-72 hours of high-dose intravenous furosemide started at the time of hospital admission, patients admitted with AHF will be randomized to open-label oral treatment with either low-dose sequential nephron blockade or high-dose furosemide for 96 hours.

The primary end-point will be the bivariate change in body weight and serum creatinine value at 96 hours since randomization. Secondary endpoints will include clinical (e.g., total change in body weight during hospitalization, change in dyspnea score at 96 hours since randomization, 30-day readmission rate) and laboratory (e.g., change in BNP or NT-proBNP at discharge vs randomization) parameters, and safety (e.g., change in serum creatinine value at discharge versus randomization and up to 30 days from discharge) issues.

DETAILED DESCRIPTION:
The SEEQUOIA-AHF trial is aimed at ascertaining if the early, oral administration of a combination of four diuretics with different sites of action along sequential nephron segments (i.e., sequential nephron blockade: proximal tubule, loop of Henle, distal tubule, cortical collecting duct) may achieve greater decrease in body weight and lower increase in serum creatinine values as compared with standard of care, i.e. a conventional diuretic therapy regimen based on high-dose oral furosemide. To assess the efficacy and safety of an early sequential nephron blockade, the study intervention will be initiated 24-72 hours after an algorithm-based treatment with high-dose intravenous furosemide started at the time of hospital admission to achieve patient stabilization.

After 24-72 hours of algorithm-based treatment with high-dose intravenous furosemide, eligible patients will be randomized to either control (furosemide-only) or intervention (early sequential nephron blockade) arm.

All patients will be put on a low sodium diet (< 70 mEq/24 hours), and will be allowed a fluid intake of < 1 L/day.

Following randomization patients will be started on oral diuretic therapy according to two different approaches, namely:

1. High-dose oral furosemide-only arm A furosemide oral dose equivalent to twice the intravenous dose of the last 24 hours will be given in two daily divided doses.

   Unless serum potassium value is higher than 5.0 mEq/L, oral spironolactone or potassium canrenoate will be added; dose will be established based on serum creatinine value Oral or intravenous potassium supplementation (potassium chloride at least 24 mEq/day) will be started if serum potassium value is lower than 4.0 mEq/L
2. Early sequential oral diuretic nephron blockade

   1. Furosemide A furosemide oral dose equivalent to the previous 24-hour intravenous dose will be given in two divided doses
   2. Metolazone. Dose will be established based on serum creatinine value
   3. Acetazolamide. Dose will be established based on serum creatinine value
   4. Spironolactone or Potassium Canrenoate. Unless serum potassium value is higher than 5.0 mEq/L, oral spironolactone or potassium canrenoate will be added; dose will be established based on serum creatinine value.

In both arms, if within the first 48 hours since randomization urine output is lower than 1.5 L/day and/or body weight decrease is less than 0.5 Kg/day, the oral dose of furosemide will be doubled, or the patient will be switched to intravenous administration at the discretion of the attending physician. If urinary output exceeds 50 ml/Kg/day current furosemide dose will be halved. Diuretics can be decreased or temporarily discontinued if there is a decrease in systolic blood pressure (> 25% of basal value) or worsening kidney function (WKF, defined as an increase in serum creatinine value ≥ 0.3 mg/dL or 25% from baseline value within 24-48 hours) that is felt as being be due to a transient episode of intravascular volume depletion. After the patient has stabilized, if congestion persists, diuretics will be reinitiated or their doses will be increased until the patient's fluid balance has been optimized. Investigators may opt-out of the treatment algorithm if they feel that it is in the interest of patient care.

The primary endpoint will be the bivariate change in body weight and serum creatinine value at 96 hours since patient randomization.

According to the data from the study of Grodin et al (J Card Fail 2016; 22:26-32), comparing subjects randomized to stepped-care diuretic treatment in the Cardiorenal Rescue Study in Acute Decompensated Heart Failure (CARRESS-HF) trial with those developing the cardiorenal syndrome during standard treatment with intravenous furosemide in the Diuretic Optimization Strategies Evaluation Acute Heart Failure (DOSE-AHF) trial and the Renal Optimization Strategies Evaluation in Acute Heart Failure (ROSE-AHF) trial, the mean difference in body weight obtained with the stepped-care oral approach versus the intravenous approach was -1.2 Kg, with a standard deviation (SD) ranging between 1.5 and 2.4 Kg; the mean difference in serum creatinine was -0.1 mg/dL, with a SD of 0.3 mg/dL. Thus, the investigators estimated that the enrollment of 206 patients would yield a 90% power to detect a 0.5 effect size for either component of the bivariate primary endpoint (1.2/2.4 Kg and 0.15/0.30 mg, respectively) with a two-sided 0.05 alpha level.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female patient, 18 years or older
* Patients admitted to Cardiology or Internal Medicine units with a diagnosis of acute decompensated heart failure and congestion: NT-proBNP > 1,000 pg/ml or BNP >250 pg/ml, dyspnea and at least two of the following clinical signs: 2+ pitting edema, pulmonary edema/pleural effusions at chest x-ray or US body weight increase above usual > 5% over the last 4 weeks
* Clinically stable patients that can be switched to oral diuretic therapy after 24-72 hours of an algorithm-based treatment with high-dose intravenous furosemide started at the time of hospital admission
* Patients capable to provide written informed consent

Exclusion Criteria:

* Serum creatinine levels > 3.5 mg per deciliter at admission to the hospital or usual estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73 m2 by the MDRD or CKD-EPI formula
* Systolic blood pressure < 90 mmHg at time of enrollment and/or hemodynamic instability severe enough to require intravenous inotropes, intravenous vasodilators, or both
* Severe arrhythmias with hemodynamic instability or DC shock occurred prior to randomization
* Ascertained acute coronary syndrome (ACS), or ACS occurred within the last 4 weeks
* Hematocrit > 45%
* Use of iodinated radio contrast material occurred in the last 72 hours
* Current mechanical ventilator support
* Previous solid organ transplant
* Primary hypertrophic or infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis or cardiac tamponade, severe valvular stenosis
* Complex congenital heart disease
* Liver disease (serum ALT or AST > 4, and/or total serum bilirubin > 3)
* Known bilateral renal artery stenosis
* Active sepsis or ongoing systemic infection
* Active gastrointestinal tract bleeding
* Enrollment in another clinical trial
* Locally advanced or metastatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Body weight change at 96 hours since randomization | 96 hours since randomization
  Difference between body weight (in Kg) at 96 hours since randomization and the value at randomization
Serum creatinine change at 96 hours since randomization | 96 hours since randomization
  Difference between the concentration of serum creatinine (in mg/dL) at 96 hours since randomization and the value at randomization

SECONDARY OUTCOMES:
Efficacy: Total weight change during hospitalization | Up to 30 days
  Difference between body weight (in Kg) at discharge and the value at admission
Efficacy: Percent change in body weight at discharge versus at randomization | Up to 30 days
  Percent change in body weight at discharge relative to the value at randomization
Efficacy: Change in dyspnea score at 96 hours since randomization | 96 hours since patient randomization
  Difference in dyspnea score (visual analog scale, VAS) at 96 hours since randomization and the score at randomization. For each patient, a plot of the respective VAS score over time will be constructed with points existing for each of the VAS measurements at pre-specified time points (e.g., randomization, 24 hours after randomizatio, etc, through 96 hours after randomization). A straight line will be drawn connecting each of the points showing the trend over time. The area under the entire piecewise line is the response variable. Increasing values indicate worse dyspnea, and viceversa. Range of VAS is approximately 0 to 900 points
Efficacy: Total equivalent furosemide dose at 96 hours since randomization | 96 hours since patient randomization
  Total equivalent furosemide dose administered within the first 96 hours since randomization
Efficacy: Proportion of patients requiring an increase in furosemide dose or switching to intravenous infusion within the first 96 hours since randomization | 96 hours since patient randomization
  Proportion of patients requiring an increase in furosemide dose or switching to intravenous infusion within the first 96 hours since randomization
Efficacy: Change in BNP or NT-pro BNP serum concentrations at discharge versus at randomization | Up to 30 days
  Difference between in BNP or NT-pro BNP serum concentrations at discharge and values at randomization
Efficacy: Percentage of patients with BNP or NT-pro BNP decrease > 30% at discharge versus at randomization | Up to 30 days
  Percentage of patients with BNP or NT-pro BNP serum concentration decrease > 30% at discharge relative to the value at randomization
Efficacy: Length-of-hospital stay | Up to 30 days
  Duration of patient hospitalization, in days
Efficacy: 30-day readmission rate | 30 days since patient discharge
  Rate of hospital readmission within 30 days since patient discharge
Safety: Change in serum creatinine value at discharge versus at randomization | Up to 30 days
  Difference between serum creatinine value (in mg/dL) at discharge and the value at randomization
Safety: Change in serum creatinine concentration at 30 days since discharge versus at randomization | Since patient randomization to 30 days after discharge
  Difference between serum creatinine concenctration at 30 days since discharge and the value at randomization
Safety: Change in BUN/creatinine ratio at 96 hours since randomization | 96 hours since randomization
  Difference between serum urea nitrogen/creatinine ratio at 96 hours since randomization and the value at randomization
Safety: Change in BUN/creatinine ratio at discharge versus at randomization | Up to 30 days
  Difference in serum urea nitrogen/creatinine ratio at discharge and the value at randomization
Safety: Change in BUN/creatinine ratio at 30 days since discharge versus at randomization | Since patient randomization to 30 days after discharge
  Difference in serum urea nitrogen/creatinine ratio at 30 days since discharge and the value at randomization
Safety: Percentage of patients with WKF at 96 hours since randomization | 96 hours since randomization
  Percentage of patients with worsening kidney function at 96 hours since randomization
Safety: Percentage of patients with WKF at discharge versus at randomization | Up to 30 days
  Percentage of patients with worsening kidney function at discharge versus at randomization
Safety: Percentage of patients with hyponatremia at 96 hours since randomization | 96 hours since randomization
  Percentage of patients with serum sodium concentration less than 136 mEq/L at 96 hours since randomization
Safety: Percentage of patients with severe hyponatremia at 96 hours since randomization | 96 hours since randomization
  Percentage of patients with serum sodium concentration lower than 125 mEq/L at 96 hours since randomization
Safety: Percentage of patients with hypernatremia at 96 hours since randomization | 96 hours since randomization
  Percentage of patients with serum sodium concentration higher than 144 mEq/L at 96 hours since randomization
Safety: Percentage of patients with hypokalemia at 96 hours since randomization | 96 hours since randomization
  Percentage of patients with serum potassium concentration lower than 3.5 mEq/L at 96 hours since randomization
Safety: Percentage of patients with hyperkalemia at 96 hours since randomization | 96 hours since randomization
  Percentage of patients with serum potassium concentration higher than 5.5 mEq/L at 96 hours since randomization
Safety: Percentage of patients with metabolic alkalosis at 96 hours since randomization | 96 hours since randomization
  Percentage of patients with plasma bicarbonate concentration higher than 30 mEq/L at 96 hours since randomization
Safety: Percentage of patients with hypomagnesemia at 96 hours since randomization | 96 hours since randomization
  Percentage of patients with serum magnesium concentration lower than 1.6 mg/dL at 96 hours since randomization
Safety: Days with hyponatremia since randomization to discharge | Up to 30 days
  Days with serum sodium concentration less than 136 mEq/L since randomization to discharge
Safety: Days with severe hyponatremia since randomization to discharge | Up to 30 days
  Days with serum sodium concentration less than 125 mEq/L since randomization to discharge
Safety: Days with hypernatremia since randomization to discharge | Up to 30 days
  Days with serum sodium concentration higher than 144 mEq/L since randomization to discharge
Safety: Days with hypokalemia since randomization to discharge | Up to 30 days
  Days with serum potassium concentration lower than 3.5 mEq/L since randomization to discharge
Safety: Days with hyperkalemia since randomization to discharge | Up to 30 days
  Days with serum potassium concentration higher than 5.5 mEq/L since randomization to discharge
Safety: Days with metabolic alkalosis since randomization to discharge | Up to 30 days
  Days with plasma bicarbonate concentration higher than 30 mEq/L since randomization to discharge
Safety: Days with hypomagnesemia since randomization to discharge | Up to 30 days
  Days with serum magnesium concentration lower than 1.6 mg/dL since randomization to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Fiaccadori, MD, PhD, Principal Investigator — Universita degli Studi di Parma; Giuseppe Regolisti, MD, Study Director — UO Nefrologia, Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- UO Nefrologia, Azienda Ospedaliero-Universitaria di Parma, Parma, PR, Italy

IPD SHARING:
Plan to Share IPD: No